CLINICAL TRIAL: NCT02649179
Title: Local Infiltration With Ropivacaine Improves Postoperative Pain Control in Patients Undergoing Laparoscopic Cholecystectomy: a Prospective, Randomized, Placebo Controlled, Double-blind Trial
Brief Title: Local Infiltration With Ropivacaine Improves Postoperative Pain Control in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Doctor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-ESR-14-10228
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local infiltration with ropivacaine (Experimental): patients were to receive 0.75% ropivacaine
  Interventions: Drug: Ropivacaine
- local infiltration with 0.9% saline (Placebo Comparator): patients were to receive placebo
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Ropivacaine — All wounds were infiltrated with 0.75% ropivacaine 14ml at port sites before wound closure(6ml for epigastric port ,6ml for umbilical port ,and 4ml for working port) . The study drugs will be applied to the skin, subcutis, fascia, and parietal peritoneum through the port sites at the end of surgery.
  Other Names: Naropin
  Arms: local infiltration with ropivacaine
Drug: 0.9% saline — All wounds were infiltrated with 0.9% saline 14ml at port sites before wound closure(6ml for epigastric port ,6ml for umbilical port ,and 4ml for working port) . The study drugs will be applied to the skin, subcutis, fascia, and parietal peritoneum through the port sites at the end of surgery.
  Other Names: saline
  Arms: local infiltration with 0.9% saline

SUMMARY:
The purpose of this study is to evaluate the effect of pain relief after infusion of ropivacaine at port sites at end of laparoscopic cholecystectomy (LC)compared with placebo (0.9% normal saline).

DETAILED DESCRIPTION:
Patients were randomly assigned to two groups, On Day 1,each subject was to undergo laparoscopic cholecystectomy under general anesthesia. Anesthesia will be induced with fentanly (2-4ug/kg), propofol TCI (4ug/ml), rocuronium (0.6mg/kg), and maintaine with remifentanly(0.1-0.3ug/kg.h) , and propofol TCI (3-5ug/ml). At the end of the operation before wound closure, patients were randomized 1:1 to receive ropivacaine or placebo. In study group all wounds were infiltrated with 0.75% ropivacaine 14ml at port sites before wound closure(6ml for epigastric port ,6ml for umbilical port ,and 4ml for working port) . The study drugs will be applied to the skin, subcutis, fascia, and parietal peritoneum through the port sites at the end of surgery. All anesthetics will be stopped when wound infiltration completed. Patients will be send to PACU for monitor a while then back to ward. Record of pain intensity evaluation and rescue analgesic medication consumption were to continue through 48hours after administration of study drug. Pain intensity will be assessed by using a 0-10 point VAS scale. VAS-rest and VAS-coughing were recorded at the baseline ,2,4,6,8,12,18,24,48 hours. Postoperative Rescue analgesia consisit of Parecoxib Sodium 40mg be given by a nurse on requst of the subject to a maximum of 80mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, and any race, Age≥18 years at the screening visite.
* ASA physical status I to II.
* Scheduled to undergo laparoscopic cholecystectomy under general anesthesia.
* Famale subjects must be without pregnancy.
* Ability to provide informed consent, adhere to the study visite schedule, and complete all study assessments.

Exclusion Criteria:

* Boss mass index >35kg/㎡
* Under intravertebral anesthesia and/or epidural analgesia
* Under postoperatived patient-controlled epidural analgesia (PCEA) and postoperative intravenous analgesia(PCIA).
* Inability to understand and use the visual analog scale (VAS)
* Currently pregnant,nursing,or planning to become pregnant during the study or within one month after study drug administration.
* Chronic user of analgesic medications, including taking opioid medications for more than 14 days in the last 3months,or non-opioid pain medications more than 5 times per week.
* Proven or suspected allergy to local anesthetics ,NSAIDs and opioids .
* Use of any NSAIDs including selective COX-2 inhibitor , opioids or other analgesic agents within 3days of surgery.
* History of suspected or known addiction to or abuse of drugs or alcohol within the past 2 years.
* Current acute or chronic medical or major psychiatric disease that,in the opinion of the investigator ,would interfere with the evaluation of study drug efficacy or safety.
* Any other subjects were not suitable to this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The area under the curve of visual analog scale (VAS) pain intensity scores at rest through 24h postoperative | 0-24h postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Lu, MD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No